CLINICAL TRIAL: NCT02707042
Title: Microbial, Immune, and Metabolic Perturbations by Antibiotics (MIME Study)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 160078; 16-I-0078
Record Dates: First submitted 2016-03-08; First posted 2016-03-14 (Estimated); Last update posted 2025-09-11 (Actual); Status verified 2025-09-09

CONDITIONS: Normal Physiology; Healthy
Keywords: Microbiome; Amoxicillin; Azithromycin; Stool; Healthy
MeSH Terms: interventions — Amoxicillin; Azithromycin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group A (Other): Control
  Interventions: Other: Control
- Group B (Other): Amoxicillin
  Interventions: Drug: Amoxicillin
- Group C (Other): Azithromycin
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Amoxicillin — 7-day therapeutic oral course of twice daily amoxicillin
  Arms: Group B
Drug: Azithromycin — 5-day oral course of once-daily azithromycin
  Arms: Group C
Other: Control — A group of volunteers will receive no antibiotics and will serve as study controls.
  Arms: Group A

SUMMARY:
More than 250 million courses of antibiotics are prescribed annually in the ambulatory care setting in the United States alone, including more than 40 million in children under 18 years of age. The perception that antibiotic use has minimal attendant adverse side effects contributes to the over-utilization of antibiotics in clinical circumstances when they are not strictly indicated. We have learned much about the human microbiome. The emerging view is of profound life-long bi-directional interactions between our microbiota and our cells. Perturbations in the microbiota affect metabolic, immune, and cognitive physiology in experimental animal models. When a person takes an antibiotic, the antibiotic diffuses via the blood into all body compartments, selecting for resistance. We propose to examine the effects of two commonly used antibiotics (the beta-lactam, amoxicillin and the macrolide azithromycin) on human microbial populations and on metabolic and immune physiology, studying healthy human volunteers in a randomized controlled clinical trial at the NIH Clinical Center. Our hypothesis is that in addition to acutely perturbing the human microbiome, these agents will have measurable metabolic and immunologic effects, with residual effects in the weeks that follow. To test this hypothesis, we will assess the effects of a brief therapeutic course of antibiotics on microbiome and metagenome composition. After an initial evaluation period, antibiotics will be given for 7 days or 5 days (depending on the antibiotic), and there will be a post-treatment evaluation. A control group will receive no drug intervention. Specimens will be obtained from multiple sites at each of 10 time points occurring before, during, and after antibiotic administration, and used for estimating bacterial and fungal composition and gene content. We will also assess the effects of the antibiotic course on markers of innate and adaptive immunity as well as markers of metabolic and hormonal physiology. A subgroup of subjects will be studied in the clinical center metabolic chamber to assess 24-hour energy expenditure and its components (sleeping, diet-induced, and activity energy expenditure), as well as macronutrient oxidation rates (carbohydrate, fat, and protein), during 3 of the 10 study visits. In addition to the primary data analyses, we will build a model that integrates the temporal data to begin to understand the complex intertwined physiology between microbiome and host.

DETAILED DESCRIPTION:
More than 250 million courses of antibiotics are prescribed annually in the ambulatory care setting in the United States alone, including more than 40 million in children under 18 years of age. The perception that antibiotic use has minimal attendant adverse side effects contributes to the over-utilization of antibiotics in clinical circumstances when they are not strictly indicated. We have learned much about the human microbiome. The emerging view is of profound life-long bi-directional interactions between our microbiota and our cells. Perturbations in the microbiota affect metabolic, immune, and cognitive physiology in experimental animal models. When a person takes an antibiotic, the antibiotic diffuses via the blood into all body compartments, selecting for resistance. We propose to examine the effects of two commonly used antibiotics (the beta-lactam, amoxicillin and the macrolide azithromycin) on human microbial populations and on metabolic and immune physiology, studying healthy human volunteers in a randomized controlled clinical trial at the NIH Clinical Center. Our hypothesis is that in addition to acutely perturbing the human microbiome, these agents will have measurable metabolic and immunologic effects, with residual effects in the weeks that follow. To test this hypothesis, we will assess the effects of a brief therapeutic course of antibiotics on microbiome and metagenome composition. After an initial evaluation period, antibiotics will be given for 7 days or 5 days (depending on the antibiotic), and there will be a post-treatment evaluation. A control group will receive no drug intervention. Specimens will be obtained from multiple sites at each of 10 time points occurring before, during, and after antibiotic administration, and used for estimating bacterial and fungal composition and gene content. We will also assess the effects of the antibiotic course on markers of innate and adaptive immunity as well as markers of metabolic and hormonal physiology. A subgroup of subjects will be studied in the Clinical Center metabolic chamber to assess 24-hour energy expenditure and its components (sleeping, diet-induced, and activity energy expenditure), as well as macronutrient oxidation rates (carbohydrate, fat, and protein), during 3 of the 10 study visits. In addition to the primary data analyses, we will build a model that integrates the temporal data to begin to understand the complex intertwined physiology between microbiome and host.

ELIGIBILITY:
* SUBJECT INCLUSION CRITERIA:

Healthy women and men will be eligible for study participation if they meet the following criteria:

* A participant will have passed his/her 18th birthday and will not have attained the age of 50 at the time of enrollment.
* Willing to allow storage of their biological samples.
* Able to comply with study procedures and swallow capsules.

SUBJECT EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from study participation:

* Body Mass Index (BMI) greater than or equal to 35 or less than or equal to 18 kg/M(2).
* Vital signs outside of acceptable range at Screening Visit, i.e., blood pressure >160/100, oral temperature >100 degrees F, pulse >100.
* Use of any of the following drugs or devices within the last 6 months:

  * systemic antibiotics, antifungals, antivirals, or antiparasitics (intravenous, intramuscular, or oral);
  * oral, intravenous, intramuscular, nasal, or inhaled corticosteroids;
  * cytokines;
  * methotrexate or immunosuppressive cytotoxic agents;
  * large doses of commercial probiotics consumed (greater than or equal to 10(8) cfu or organisms per day), including tablets, capsules, lozenges, chewing gum, or powders in which probiotic is a primary component. Ordinary dietary components such as fermented beverages/milks, yogurts, and foods do not apply.
  * anabolic steroids;
  * intrauterine device, combination hormone vaginal ring for contraception (due to unknown duration of local hormone effects), topical or systemic estrogens. Oral contraceptives with a standard 28-day cycle will be permitted if the subject has been consistently taking them for at least 1 month;
  * oral, topical, intramuscular testosterone preparations.
* Illicit drug use, including amphetamines, cocaine, or heroin, within the last 6 months. Marijuana use is not exclusionary.
* Chronic smokers and subjects who use smokeless tobacco products (due to known effects of tobacco on the oral microbiome).
* Claustrophobia.
* Use of antacids (proton pump inhibitors, sucralfate, H1 and H2 antagonists, and those containing aluminum magnesium) within the last 3 months.
* Use of laxatives or enemas within the last 3 months.
* Diagnostic colonoscopy within the last 6 months.
* Use of topical antibiotics or topical steroids on the face, scalp, or neck, or on arms, forearms, or hands within the previous 30 days.
* Use of vaginal/vulvar medications, including antifungals, within the previous 30 days. Subjects may continue to use permitted vaginal contraceptives (spermicides and female condoms) until 24 hours prior to sampling
* Use of isotretinoin within the past 5 years.
* Intranasal influenza vaccination within the last 6 months due to effects on mucosal immunity.
* Acute disease at the time of enrollment (defer enrollment until subject recovers). Acute disease is defined as the presence of a moderate or severe illness with or without fever.
* Chronic, clinically significant (unresolved, requiring ongoing medical management or medication) pulmonary, cardiovascular, dermatologic, endocrine, GI, hepatic, or renal functional abnormality, as determined by medical history, physical examination, and/or laboratory testing. Includes, but not limited to:

  * A history of diabetes mellitus (Type 1 or 2), pituitary disease, hypothyroidism, hyperthyroidism
  * A history of physician-diagnosed asthma
  * A history of allergy to any antibiotic medications, including amoxicillin (penicillin) and/or azithromycin (macrolide)
  * A history of food allergy requiring dietary accommodation
  * Lactose-intolerance requiring dietary accommodation
  * A history of a bleeding disorder
  * Mononucleosis
  * Liver disease, including non-alcoholic fatty liver disease, AST or ALT > 1.5 times normal value, cirrhosis
  * Renal disease, as defined by serum creatinine concentrations > 1.5 mg/dL and/or overt proteinuria
  * Central nervous system disease, including previous history of cerebrovascular accidents, dementia, and neurodegenerative disorders
  * Clinically significant abnormal results on electrocardiogram (ECG) that in the opinion of the PI, would place the patient at increased risk of QT-prolongation or other cardiac event
* Genitourinary/Gynecologic conditions, including:

  * Treatment for or suspicion of ever having had toxic shock syndrome
  * History of hysterectomy or oophorectomy
  * History of condyloma or human papillomavirus diagnosed within the previous 2 years
  * History of candidiasis, urinary tract infection, or sexually transmitted disease (specifically chlamydia, gonorrhea, syphilis, genital herpes, trichomoniasis) diagnosed within the previous 6 months
  * Evidence (by history or physical exam) of vulvar or vaginal irritation at screening
  * History of vulvar, vaginal, or cervical dysplasia within the previous 5 years
* History of cancer except for squamous or basal cell carcinomas of the skin that have been medically managed by local excision.
* Unstable dietary history as defined by major changes in diet during the previous month, where the subject has eliminated or significantly increased a major food group in the diet.
* Recent history of excessive alcohol consumption defined as more than five 1.5-ounce servings of 80-proof distilled spirits, five 12-ounce servings of beer, or five 5-ounce servings of wine at one sitting over the last 30 days.
* Positive test for HIV, hepatitis B virus, or hepatitis C virus indicating infection (hepatitis B seropositivity conferred by vaccination is not exclusionary).
* Any confirmed or suspected condition/state of immunosuppression or immunodeficiency (primary or acquired).
* Major surgery of the GI tract, including cholecystectomy or appendectomy, in the past 5 years. Any major bowel resection at any time.
* History of gastric stapling, lap band, or surgical procedure for treatment of obesity.
* History of GI disorders or diseases including:

  * inflammatory bowel disease (IBD) including ulcerative colitis, Crohn s disease (of any severity), or indeterminate colitis;
  * irritable bowel syndrome (IBS);
  * persistent, infectious gastroenteritis, colitis or gastritis, persistent or chronic diarrhea of unknown etiology, Clostridium difficile infection (recurrent), gastric or duodenal ulcer;
  * Celiac disease;
  * chronic constipation.
* Active behavioral or psychiatric conditions that would be incompatible with a safe and successful participation in the study, including major depression, anxiety disorder, schizophrenia, and presence of psychotic symptoms.
* Active eating disorders, including anorexia nervosa, bulimia, or binge eating syndrome.
* Use of weight-loss drugs within the past 5 years.
* Weight change (intended or unintended; loss or gain) of more than 10% of total body weight in the 3 months before admission.
* Regular urinary incontinence necessitating use of incontinence protection garments.
* Female who is pregnant, intending to become pregnant, or lactating.
* History of recurrent rashes within the past 6 months.
* At the time of the screening visit:

  * multiple blisters, pustules, boils, abscesses, erosions or ulcers on the scalp, face, neck, arms, forearms, or hands;
  * uniformly thickened, cracking, dry skin on bilateral palms and/or soles;
  * disseminated rash (at multiple body sites or extending throughout a broad body area).
* Subjects who are unable to complete required study visits per allotted visit windows.
* Any condition that, in the opinion of the investigator, contraindicates participation in this study.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2017-03-22 (Actual); Primary Completion 2025-05-14 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
To determine whether antibiotic-induced perturbation of the microbiome has measurable metabolic and immunologic effects during and after the treatment period. | Prior to, during, after antibiotic course
  1. Change in total EE of 5% from pre-treatment to post-treatment among the subjects receiving antibiotics (metabolic endpoint). 2. Average decrease of 500 cell/mm3 in the peripheral blood leukocyte count from pre-treatment to post-treatment among subjects receiving antibiotics (immunologic endpoint).

SECONDARY OUTCOMES:
Changes in parameters of metabolic functioning, including measures of hormones relevant to metabolism. | Prior to, during, after antibiotic course
  Changes in 24-hr EE, its components (sleeping, diet-induced, and activity EE), macronutrient oxidation rates (carbohydrate, fat, and protein), core body temperature (to evaluate circadian rhythm), and heart rate variability (as a measure of sympathetic versus parasympathetic nervous system activities).
Changes in blood, cutaneous, intestinal, oral, salivary, urinary, vaginal bacterial microbiomes; | Prior to, during, after antibiotic course
  Alterations in relative abundance and function of peripheral blood cells and specialized subsets as they relate to innate and adaptive immune pathways.
Changes in parameters of immune function and response in samples of blood, serum/plasma; and | Prior to, during, after antibiotic course
  Changes in markers of innate and adaptive immunity as detected in serum, urine, saliva and feces, which may include immunoglobulins, cytokines, chemokines, markers of bacterial translocation and markers of systemic and mucosal inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Christa S Zerbe, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McCaig LF, Besser RE, Hughes JM. Antimicrobial drug prescription in ambulatory care settings, United States, 1992-2000. Emerg Infect Dis. 2003 Apr;9(4):432-7. doi: 10.3201/eid0904.020268. PMID 12702222
- [Background] McCaig LF, Hughes JM. Trends in antimicrobial drug prescribing among office-based physicians in the United States. JAMA. 1995 Jan 18;273(3):214-9. PMID 7807660
- [Background] Grijalva CG, Nuorti JP, Griffin MR. Antibiotic prescription rates for acute respiratory tract infections in US ambulatory settings. JAMA. 2009 Aug 19;302(7):758-66. doi: 10.1001/jama.2009.1163. PMID 19690308
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-I-0078.html